CLINICAL TRIAL: NCT02130804
Title: Using Salsalate to Target Adipocyte Macrophage Infiltration and Reverse Metabolic Disease Risk in Obese Hispanic Young Adults
Brief Title: Using Salsalate to Target Adipocyte Macrophage Infiltration
Acronym: TAMI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Michael I. Goran, Professor in the Departments of Preventive Medicine, Physiology & Biophysics and Pediatrics in the Keck School of Medicine, Director of the Childhood Obesity Research Center, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HS-11-00017
Record Dates: First submitted 2014-04-29; First posted 2014-05-05 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Risk
Keywords: Obesity; Adipose tissue inflammation; Salsalate; Hispanics
MeSH Terms: conditions — Obesity | interventions — salicylsalicylic acid; Salicylates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Salsalate (Experimental): Salsalate (4 g/day)
  Interventions: Drug: Salsalate (4 g/day)
- Placebo (Placebo Comparator): Placebo (4 g/day)
  Interventions: Drug: Placebo (4 g/day)

INTERVENTIONS:
Drug: Salsalate (4 g/day) — Given orally twice daily
  Other Names: Salicylate
  Arms: Salsalate
Drug: Placebo (4 g/day) — Given orally twice daily
  Other Names: Inactive control
  Arms: Placebo

SUMMARY:
Background: The prevalence of obesity has increased throughout the last three decades due to genetic, metabolic, behavioral, and environmental factors. Obesity and high-fat western diets activate inflammatory processes, which promote development of insulin resistance as well as other metabolic complications. Increasing obesity rates are a major public health concern in the Hispanic population due to the large number of Hispanics suffering from obesity. Based on preliminary data, we propose a double-blind randomized clinical trial of Salsalate therapy in obese Hispanic young adults. Salsalate treatment shows promise for decreasing inflammation under conditions of weight stability by reducing macrophage infiltration of adipocytes. Hispanics have the greatest amount of visceral adipose tissue (VAT), liver fat, and inflammation when compared to other ethnic groups, thereby increasing the potential for treatment effects in this high-risk population.

Purpose: The purpose of this study is to demonstrate through a "proof-of-concept" trial that Salsalate induced reductions in adipose tissue inflammation are possible under conditions of weight stability.

Methodology: We will recruit obese Hispanic young adults (18 - 35 years) from hospitals, clinics, and community centers. Study Endpoints: Primary outcomes will be macrophage infiltration as assessed by the presence of crown-like structures (CLS) in subcutaneous adipose tissue (SAT) biopsies, liver fat, insulin sensitivity, and fasting glucose. We will also assess plasma levels of monocyte chemoattractant protein (MCP)-1, tumor necrosis factor (TNF)-α, interleukin (IL)-1, C-reactive protein (CRP), and SAT gene expression of nuclear factor kB (NF-kB) and insulin signaling pathways.

Intervention and Follow-up: Participants will be randomly assigned to four weeks of treatment with Salsalate (4 g/d) or placebo and will be studied under weight maintenance conditions. These measures will enable us to determine if Salsalate treatment is capable of reducing adipose tissue inflammation and related metabolic outcomes in the absence of weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Obese (body mass index >30 kg/m^2)
* Hispanic males and females age 18-35 years

Exclusion Criteria:

* Women with hemoglobin <11.5 g/dL or men with hemoglobin <12.5 g/dL will be excluded
* AST / ALT >2 times the upper limit of normal
* Evidence of any liver disease other than non-alcoholic steatosis
* Diabetes
* Diagnosis of any disease that is known to influence insulin action and secretion
* Current or past involvement in any weight loss, exercise, or sports program in the six months prior to participation
* Use of medication known to influence body composition or fat distribution (e.g. Cushing syndrome)
* History of renal disease
* Use of non-steroidal anti-inflammatory drugs (NSAIDs)
* Chicken pox, flu, or influenza infection
* Those taking high doses of vitamin C, antacids (containing Ca2+ or Mg+2), or taking Warfarin
* Hypertension
* Allergies to Salsalate, aspirin or other NSAIDs
* History of peptic ulcer or upper GI bleeding
* A positive pregnancy test or current lactation
* Has smoked greater than 100 cigarettes in their lifetime and now smokes everyday or some days
* Drinks greater than 200 g/day of alcohol
* Those with a waist circumference (or widest part of body measurement) greater than or equal to 185 cm due to MRI size restrictions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in plasma glucose levels over a 2-hour oral glucose tolerance test | 4 weeks
  Glucose following 4 weeks of treatment with salsalate (4 g/day) or placebo. A 2-hour oral glucose tolerance test will be performed at baseline and 4 weeks to measure changes in plasma glucose levels.
Change in adipose tissue inflammation | 4 weeks
  Adipose tissue inflammation following 4 weeks of treatment with salsalate (4 g/day) or placebo. Adipose tissue inflammation will be determined from abdominal subcutaneous adipose tissue biopsies performed at baseline and 4 weeks.
Change in systemic markers of inflammation | 4 weeks
  Systemic markers of inflammation following treatment with salsalate (4 g/day) or placebo. Fasting blood samples will be taken at baseline and 4 weeks to measure systemic markers of inflammation.
Change in plasma insulin levels over a 2-hour oral glucose tolerance test | 4 weeks
  Insulin following 4 weeks of treatment with salsalate (4 g/day) or placebo. A 2-hour oral glucose tolerance test will be performed at baseline and 4 weeks to measure changes in plasma insulin levels.
Change in plasma fasting free fatty acid levels | 4 weeks
  Fasting free fatty acids (FFA) following 4 weeks of treatment with salsalate (4 g/day) or placebo. Fasting blood samples will be taken at baseline and 4 weeks to measure changes in plasma fasting FFA.
Change in plasma C-peptide levels over a 2-hour oral glucose tolerance test | 4 weeks
  C-peptide following 4 weeks of treatment with salsalate (4 g/day) or placebo. A 2-hour oral glucose tolerance test will be performed at baseline and 4 weeks to measure changes in plasma C-peptide levels.

SECONDARY OUTCOMES:
Change in body composition | 4 weeks
  Changes in body composition following 4 weeks of treatment with salsalate (4 g/day) or placebo. A DEXA scan will be performed at baseline and 4 weeks to measure any potential changes in body composition (body fat and lean tissue mass).
Change in ectopic fat | 4 weeks
  Changes in ectopic fat following 4 weeks of treatment with salsalate (4 g/day) or placebo. A 3-Tesla whole abdominal MRI scan will be performed at baseline and 4 weeks to measure any potential changes in ectopic fat.
Change in diet | 4 weeks
  Changes in diet following 4 weeks of treatment with salsalate (4 g/day) or placebo. A 24-hour diet recall will be performed at baseline and 4 weeks to measure any potential changes in diet.
Change in physical activity | 4 weeks
  Changes in physical activity following 4 weeks of treatment with salsalate (4 g/day) or placebo. A Godin-Shephard Leisure-Time Physical Activity questionnaire will be performed at baseline and 4 weeks to measure any potential changes in physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Michael I Goran, PhD, Principal Investigator — University of Southern California; Tanya L Alderete, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - University of Southern California Diabetes Obesity Research Institute (DORI), Los Angeles, California
  - University of Southern California, Clinical Trials Unit (CTU), Los Angeles, California

REFERENCES:
- [Background] Goldfine AB, Conlin PR, Halperin F, Koska J, Permana P, Schwenke D, Shoelson SE, Reaven PD. A randomised trial of salsalate for insulin resistance and cardiovascular risk factors in persons with abnormal glucose tolerance. Diabetologia. 2013 Apr;56(4):714-23. doi: 10.1007/s00125-012-2819-3. Epub 2013 Jan 31. PMID 23370525
- [Background] Goldfine AB, Fonseca V, Jablonski KA, Pyle L, Staten MA, Shoelson SE; TINSAL-T2D (Targeting Inflammation Using Salsalate in Type 2 Diabetes) Study Team. The effects of salsalate on glycemic control in patients with type 2 diabetes: a randomized trial. Ann Intern Med. 2010 Mar 16;152(6):346-57. doi: 10.7326/0003-4819-152-6-201003160-00004. PMID 20231565
- [Background] Goldfine AB, Silver R, Aldhahi W, Cai D, Tatro E, Lee J, Shoelson SE. Use of salsalate to target inflammation in the treatment of insulin resistance and type 2 diabetes. Clin Transl Sci. 2008 May;1(1):36-43. doi: 10.1111/j.1752-8062.2008.00026.x. PMID 19337387
- [Background] Fleischman A, Shoelson SE, Bernier R, Goldfine AB. Salsalate improves glycemia and inflammatory parameters in obese young adults. Diabetes Care. 2008 Feb;31(2):289-94. doi: 10.2337/dc07-1338. Epub 2007 Oct 24. PMID 17959861
- [Background] Koska J, Ortega E, Bunt JC, Gasser A, Impson J, Hanson RL, Forbes J, de Courten B, Krakoff J. The effect of salsalate on insulin action and glucose tolerance in obese non-diabetic patients: results of a randomised double-blind placebo-controlled study. Diabetologia. 2009 Mar;52(3):385-93. doi: 10.1007/s00125-008-1239-x. Epub 2008 Dec 23. PMID 19104769
- [Background] Faghihimani E, Aminorroaya A, Rezvanian H, Adibi P, Ismail-Beigi F, Amini M. Reduction of insulin resistance and plasma glucose level by salsalate treatment in persons with prediabetes. Endocr Pract. 2012 Nov-Dec;18(6):826-33. doi: 10.4158/EP12064.OR. PMID 22784842
- [Background] Faghihimani E, Aminorroaya A, Rezvanian H, Adibi P, Ismail-Beigi F, Amini M. Salsalate improves glycemic control in patients with newly diagnosed type 2 diabetes. Acta Diabetol. 2013 Aug;50(4):537-43. doi: 10.1007/s00592-011-0329-2. Epub 2011 Sep 22. PMID 21938543